CLINICAL TRIAL: NCT01775696
Title: The Role of Central and Systemic Inflammation and Aβ-specific Immune Responses in Early AD
Brief Title: Central and Systemic Inflammation in Alzheimer's Disease
Acronym: IMABio3
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P100145
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Pittsburgh binding Compound (PiB); Positron Emission Tomography (PET); Inflammation; Anti Abeta immune responses; Blood markers; MRI
MeSH Terms: conditions — Alzheimer Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- sporadic AD: 80 sporadic AD patients (40 at the stage of MCI, 40 at the stage of mild or moderate dementia)
- familial forms of AD: 15 familial forms of AD caused by APP, PSEN1 or PSEN2 mutations
- asymptomatic relatives: 30 asymptomatic relatives to familial AD patients
- controls: 40 controls
- genetic FTD: 5 genetic forms of FTD

SUMMARY:
The main objective of this study is to investigate the central and peripheral inflammatory, as well as the spontaneous Aβ-specific, immune responses at the asymptomatic stage and early stages of AD by combining molecular imaging techniques with blood biomarker analyses. The early and preclinical stages of AD will be studied in the relatives of patients with PSEN1, PSEN2 or APP mutations that are at-risk (50%) to be mutation carriers. This study will evaluate the contribution of Inflammatory and immune anti-Aβ responses (I2ARs) in AD progression. Inclusion of sporadic and familial forms of AD will aid in studying the chronology of pathological events. Clinical follow-ups will be conducted annually for two years and will include an MRI and a blood draw on the last visit. We expect I2ARs to appear in the early stages of the disease and to constitute new prognostic factors. I2ARs could also become therapeutic markers for the assessment of novel anti-amyloid treatments and may offer new insights to the development of Aβ-specific immunotherapy strategies.

DETAILED DESCRIPTION:
Introduction: Alzheimer's disease (AD) is characterized by abnormal β-amyloid deposition associated with Tau-based neurofibrillary tangles. The metabolism of these proteins is modulated by the individuals physiological background. In addition to genetic factors, early brain inflammation and the presence of a spontaneous beta amyloid (Aβ)-specific immune response are likely to have an important influence on amyloid pathogenesis, as demonstrated in recent neuropathological and experimental studies. In vivo measurements of the β-amyloid load and brain inflammation have become available with the development of new tracers for positron emission tomography (PET) imaging. So far, tracers for brain inflammation have had a limited ability to detect changes in the expression of peripheral benzodiazepine receptors (PBR), which are mainly present on the surface of activated microglial cells. The recently developed [18F]DPA-714 was found to be a better ligand for PBR than previous tracers. Inflammatory and immune anti-Aβ responses (I2ARs) are likely to occur very early in the pathogenic protein cascade. They could thus constitute early markers for AD diagnosis and also play key roles in its phenotypic presentation and as prognostics. Comparing sporadic AD and familial forms of AD caused by APP, PSEN1 or PSEN2 mutations (in both symptomatic and at-risk non-symptomatic relatives) will aid in establishing the chronology of pathological events and defining their clinical impact.

The main objective of this study is to investigate the central and peripheral inflammatory, as well as the spontaneous Aβ-specific, immune responses at the asymptomatic stage and early stages of AD by combining molecular imaging techniques with blood biomarker analyses. The early and preclinical stages of AD will be studied in the relatives of patients with PSEN1, PSEN2 or APP mutations that are at-risk (50%) to be mutation carriers.

The secondary objectives are

1. to investigate the specificity of the central inflammatory response (DPA PET scan) and the peripheral I2AR (blood markers) by analyzing their correlation with amyloid-binding radiotracer (PIB PET scan);
2. to evaluate the prognostic value of central and peripheral I2ARs on disease evolution over a 2 year follow-up;
3. to compare central and peripheral I2ARs in sporadic and genetic cases of AD;
4. to correlate the initial amyloid load with disease evolution in sporadic and genetic cases of AD
5. to correlate I2AR biomarkers with CSF biomarkers (Aβ1-42, tau and phosphorylated tau) when consent for lumbar puncture is obtained (optional). Each patient will then be invited to participate in a long-term follow-up study and will be informed of the possibility of brain donation for research purposes. A library of blood samples will also be collected and stored at the Platform for Biological Resources at the Salpetriere Hospital, to allow for future collaborations on new diagnostic and prognostic biomarkers based on novel techniques.

Methodology : We propose to conduct a multimodal study, first transversal, then longitudinal with a two year follow-up, based on

1. molecular PET imaging by coupling [18F]DPA-714, a marker of central inflammation, and PIB, a marker of amyloid deposition;
2. peripheral I2AR analysis (blood markers);
3. analysis of genetic factors;
4. measurement of regional cortical atrophy by MRI. A group of patients at an early stage of AD (CDR = 0.5), defined by a new diagnostic criteria (Dubois et al, 2007), will be compared to a group of moderate AD patients as defined by the criteria of NINCDS AIREN (CDR = 1 or 2), a group of patients with another type dementia (frontotemporal dementia) and a control group.

Recruitment of sporadic AD patients and controls will occur at the Pitie-Salpetriere Hospital. Teams of geneticists from Paris and Rouen will recruit patients with known mutations and at-risk asymptomatic first-degree relatives. Every subject will undergo the following examinations: (a) at the Pitie-Salpetriere Hospital, a clinical and neuropsychological assessment, a 3T multimodal research MRI, and a blood draw 8 for studying a panel of plasmatic markers, measuring the blood level of anti-Aβ antibodies, evaluating Aβ-specific T lymphocyte responses and studying potential genetic modifiers; and (b) at the ORSAY Hospital, two PET scans will be performed on the same day: first an [11C]-PIB PET scan, followed 3 hours later by an [18F]DPA-714 imaging. Clinical follow-ups will be conducted annually for two years and will include an MRI and a blood draw on the last visit.

The previous study BIOMAGE, funded by the French National Research Agency (ANR 2007), has demonstrated the logistical feasibility of the project as well as the efficiency of patient and control recruitment. The subjects that were included in BIOMAGE will be invited to participate in this research project, thus utilizing this cohort for DPA imaging and I2AR markers. The duration of the research will be four years.

Expected results and perspectives: This study will evaluate the contribution of I2ARs in AD progression. Inclusion of sporadic and familial forms of AD will aid in studying the chronology of pathological events. We expect I2ARs to appear in the early stages of the disease and to constitute new prognostic factors. I2ARs could also become therapeutic markers for the assessment of novel anti-amyloid treatments and may offer new insights to the development of Aβ-specific immunotherapy strategies.

ELIGIBILITY:
Inclusion criteria :

Sporadic AD patients at a prodromal stage:

* Be older than 30 years old.
* Progressive amnestic syndrome of the hippocampal type, defined by a free recall score

  ≤ 18 and a total recall score ≤ 40 on the Free and Cued Selective Recall Reminding Test (FCSRT).
* Absence of overt dementia.
* CDR (Clinical Dementia Rating Scale) = 0.5.
* No impact on activities of daily living, or only one item impaired at the first level of the Instrumental Activity of Daily Living Scale.
* Absence of general or systemic disorders that may interfere with cognition.
* Absence of brain lesions as determined by MRI that may account for part of the clinical presentation.

Sporadic AD patients at a mild to moderate dementia stage:

* Be older than 30 years old.
* NINCDS-AIREN criteria.
* CDR (Clinical Dementia Rating Scale) = 1 or 2

Normal controls :

* Be older than 30 years old.
* An absence of psychiatric disorder
* An absence of subjective problems with memory and normal scores on the Mini Mental State Examination (MMSE ≥ 27)

Familial symptomatic AD patients with PSEN1, PSEN2 or APP mutations:

* Be older than 18 years old.
* Patients will be identified by the team of neurogeneticists

Relatives at 50% risk of familial AD:

* These subjects will be recruited from families affected with autosomal dominant AD that is due to the mutation of the PSEN1, PSEN2 or APP genes. In these families, the first-degree relatives of patients with a mutation have a 50% risk of having the mutation that was identified in the family.

Familial frontotemporal dementia (FTD) patients :

* FTD patients with mutations in the progranulin gene or MAPT (tau) gene will be identified by the team of neurogeneticists at Rouen and Paris (Salpetriere). Familial FTD patients with known pathologies will be included regardless of the severity of the disease, given the small number of patients involved.

Concomitant therapy :

* All subjects will be asked about their history of benzodiazepine treatment: flunitrazepam, triazolam, and diazepam, which have a moderate affinity for PBR, will be forbidden or will be stopped before inclusion. Clonazepam, lorazepam, zolpidem, and zopiclone, which have a very low affinity for PBR, will be allowed. For all other benzodiazepines, specific research on their affinity toward PBR will be performed before definitive inclusion.

Subjects taking acetylcholinesterase inhibitor or memantine will be admitted.

Exclusion criteria :

* Psychiatric disorder or major depression
* Contraindication for MRI examination : carrying a cardiac pacemaker, any ferromagnetic metallic implants or foreign bodies (an internal electrical or magnetic device, a valvular prosthesis), claustrophobic subject
* Alcoholism
* Vascular lesions on MRI
* Allergy either to PiB or to DPA
* Non health insurance affiliation
* Pregnant women

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 sporadic AD patients (40 at the stage of MCI, 40 at the stage of mild or moderate dementia), 15 familial forms of AD caused by APP, PSEN1 or PSEN2 mutations, 30 asymptomatic relatives to familial AD patients, 40 controls, 5 genetic forms of FTD
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
evolution of blood markers | from 0 to 24 months
  I2AR measures [Time Frame: at 0, 12 months and 24 months]

SECONDARY OUTCOMES:
Patient's blood cell modification assessment | from M0 to M24
  Patient's blood cell modification assessment [ Time Frame: at 0, 12 months and 24 months ]
[F18] DPA-714 PET examination | Month 3
  * [F18] DPA-714 PET examination
  * Relationship between PIB examination and I2AR measures
  * Relationship between PIB examination and DPA PET examination

OTHER OUTCOMES:
Analysis of prognostic value of I2AR measures on clinical measures | 12 months
Analysis of prognostic value of I2AR measures on clinical measures | 24 months
Analysis of prognostic value of I2AR measures on neuropsychological measures | 12 months
Analysis of prognostic value of I2AR measures on neuropsychological measures | 24 months
Analysis of prognostic value of I2AR measures on hippocampal volumes | 24 months
Analysis of prognostic value of I2AR measures on hippocampal volumes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sarazin, MD, PhD, Principal Investigator — APHP
Locations (1):
- APHP - Pitié Salpetriere Hospital, Paris, France

REFERENCES:
- [Result] Corlier F, Rivals I, Lagarde J, Hamelin L, Corne H, Dauphinot L, Ando K, Cossec JC, Fontaine G, Dorothee G, Malaplate-Armand C, Olivier JL, Dubois B, Bottlaender M, Duyckaerts C, Sarazin M, Potier MC; Clinical ImaBio3 Team. Modifications of the endosomal compartment in peripheral blood mononuclear cells and fibroblasts from Alzheimer's disease patients. Transl Psychiatry. 2015 Jul 7;5(7):e595. doi: 10.1038/tp.2015.87. PMID 26151923
- [Result] Hamelin L, Bertoux M, Bottlaender M, Corne H, Lagarde J, Hahn V, Mangin JF, Dubois B, Chupin M, de Souza LC, Colliot O, Sarazin M. Sulcal morphology as a new imaging marker for the diagnosis of early onset Alzheimer's disease. Neurobiol Aging. 2015 Nov;36(11):2932-2939. doi: 10.1016/j.neurobiolaging.2015.04.019. Epub 2015 Jul 15. PMID 26256787
- [Result] Hamelin L, Lagarde J, Dorothee G, Leroy C, Labit M, Comley RA, de Souza LC, Corne H, Dauphinot L, Bertoux M, Dubois B, Gervais P, Colliot O, Potier MC, Bottlaender M, Sarazin M; Clinical IMABio3 team. Early and protective microglial activation in Alzheimer's disease: a prospective study using 18F-DPA-714 PET imaging. Brain. 2016 Apr;139(Pt 4):1252-64. doi: 10.1093/brain/aww017. Epub 2016 Mar 15. PMID 26984188
- [Derived] Peyronneau MA, Kuhnast B, Nguyen DL, Jego B, Sayet G, Caille F, Lavisse S, Gervais P, Stankoff B, Sarazin M, Remy P, Bouilleret V, Leroy C, Bottlaender M. [18F]DPA-714: Effect of co-medications, age, sex, BMI and TSPO polymorphism on the human plasma input function. Eur J Nucl Med Mol Imaging. 2023 Sep;50(11):3251-3264. doi: 10.1007/s00259-023-06286-1. Epub 2023 Jun 9. PMID 37291448